CLINICAL TRIAL: NCT00158704
Title: An Open-Label, Continued Access Study of Adefovir Dipivoxil for Patients With Chronic HBV Infection Who Have Completed a Gilead-Sponsored Study of Adefovir Dipivoxil.
Brief Title: Continued Access Study of Adefovir Dipivoxil (ADV) for Patients w/Chronic HBV Infection.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped due to marketing approval by the FDA.
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: GS-00-480
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-03-08 (Estimated); Status verified 2006-04

CONDITIONS: Hepatitis B
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — adefovir dipivoxil

INTERVENTIONS:
Drug: Hepsera

SUMMARY:
Provide adefovir dipivoxil (Hepsera) 10 mg once daily to patients with chronic hepatitis B virus (HBV) infection who have completed a Gilead-sponsored study of adefovir dipivoxil and require continued access to adefovir dipivoxil.

DETAILED DESCRIPTION:
The objective of this study is to provide adefovir dipivoxil 10 mg once daily to patients with chronic hepatitis B virus(HBV) infection who have completed a Gilead-sponsored study of adefovir dipivoxil and require continued access to adefovir dipivoxil. The secondary objective of this study is to evaluate the safety of chronic therapy with adefovir dipivoxil 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed one of the following Gilead-sponsored studies as indicated: GS-96-412, GS-98-437, GS-98-438, GS-00-461 and GS-00-481. If the patient has participated in another Gilead-sponsored study, the CRO or Sponsor's Medical Monitor will evaluate for participation in this study on a case by case basis.

Exclusion Criteria:

* Any serious or active medical or psychiatric illness that would interfere with patient treatment, assessment or compliance with the protocol or dosing requirements.
* Currently receiving nephrotoxic drugs such as aminoglycosides (e.g. amikacin, gentamicin, kanamycin, neomycin, netilmicin, streptomycin, tobramycin), amphotericin B, vancomycin, cidofovir, foscarnet, cisplatin, or pentamidine OR competitors of renal excretion such as probenecid and sulfinpyrazone. These agents must be discontinued at least 7 days prior to starting treatment with adefovir dipivoxil.
* Currently receiving investigational agents with activity against hepatitis B virus.
* Hypersensitivity to any of the components of the drug product.
* Pregnant or lactating females.
* Inability to comply with study requirements.
* Experienced a treatment limiting toxicity of adefovir dipivoxil that has not yet resolved or resulted in permanent discontinuation of adefovir dipivoxil in the previous study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2002-01; Study Completion 2005-01

PRIMARY OUTCOMES:
To provide adefovir dipivoxil (ADV) 10 mg once daily to patients with chronic hepatitis B virus (HBV) infection who have completed a Gilead-sponsored study and require continued access to ADV.

SECONDARY OUTCOMES:
To evaluate the safety of chronic therapy with ADV 10 mg.

REFERENCES:
- See also: Website for Gilead — http://www.Gilead.com